CLINICAL TRIAL: NCT04098601
Title: Inpatient Link to Addiction Recovery- a Pilot Program
Brief Title: Inpatient Link to Addiction Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Collaborators: Clemson University (Other); University of South Carolina School of Medicine, Greenville (Unknown)
Responsible Party: Principal Investigator, Prerana Roth, Clinical Assistant Professor, Prisma Health-Upstate
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00075538
Record Dates: First submitted 2019-06-11; First posted 2019-09-23 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2020-05

CONDITIONS: Substance Use Disorders
Keywords: recovery coaching; substance abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The investigator/study personnel inform the participant regarding which arm they have been assigned and inform a recovery coach if the participant is randomized to the intervention arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Recovery Coach Intervention (Experimental): Participants randomized to the intervention arm are linked to a recovery peer coach while they are in the hospital. Recovery peer coaches are provided to the participant by Faces and Voices of Recovery (FAVOR) - Greenville. Recovery coaches are Certified Peer Support Specialists (CPSS), individuals who have firsthand experience in successful recovery and are trained in using recovery-oriented tools to help peers overcome addiction. FAVOR offers immediate access to a personal coach, a local center, and assistance to off-site intervention and recovery resources in the community. They provide twice weekly contact with participants.
  Interventions: Behavioral: Recovery Coach Intervention
- Standard of Care Control (No Intervention): Patients in the control condition receive the current standard of care, which entails a treatment referral with a list of addiction recovery facilities, groups, and resources. It is the patient's responsibility to call a treatment facility or group on the list and thus relies on self-referral. The medical team is not permitted to call a facility or group on behalf of the patient. The physician may counsel the patient on the dangers of substance abuse and addiction, but the extent of counseling is variable and dependent on the individual physician.

INTERVENTIONS:
Behavioral: Recovery Coach Intervention — Participants randomized to the intervention arm are linked to a recovery peer coach while they are in the hospital. Recovery peer coaches are provided to the participant by Faces and Voices of Recovery (FAVOR) - Greenville. Recovery coaches are Certified Peer Support Specialists (CPSS), individuals who have firsthand experience in successful recovery and are trained in using recovery-oriented tools to help peers overcome addiction. FAVOR offers immediate access to a personal coach, a local center, and assistance to off-site intervention and recovery resources in the community. They provide twice weekly contact with participants.
  Arms: Recovery Coach Intervention

SUMMARY:
The objective of this proposal is to link inpatients to a certified peer support specialist through FAVOR-Greenville and determine the effectiveness of recovery coaching on patient outcomes.This study will evaluate the impact of initiating peer recovery coaching during SUD patients' hospitalization on engagement in recovery services, addiction severity, and quality of life compared to the current standard of care.

DETAILED DESCRIPTION:
The United States is in the midst of a drug overdose crisis: the rate of substance use, overdose, and substance abuse-related economic costs is rapidly increasing. Despite the prevalence of Substance Abuse Disorder (SUD), only 10% of SUD patients receive treatment. The initial link into care is often one of the hardest barriers to overcome due to wait times, complex systems to navigate, and fluctuating motivation. Hospitalization is often a time when patients are more receptive to SUD treatment. One potential effective treatment approach is peer recovery support services. Currently at Greenville Memorial Hospital, there is no direct link between hospitalization and outpatient care for patients with SUD, making it difficult to start or continue the recovery process. Thus, the goal of this study is to evaluate the impact of the initiation of peer recovery services during hospitalization on addiction severity and quality of life. By establishing a successful inpatient link to recovery treatment, this study may lead to the development of an effective method of care that can readily be implemented into the healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* English speaking;
* Identified by healthcare provider as having Substance Use Disorder
* Recent substance use
* Currently admitted to the Medical Teaching Services, general medicine hospitalist services, or Infectious Disease Consult service at Greenville Memorial Hospital

Exclusion Criteria:

* Are unable to provide informed consent (intubation, confusion, etc.) during hospitalization
* Are admitted for marijuana use only
* Are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Change in Engagement in Recovery Services | intervals of 1, 2, 3, and 6 months post-baseline assessment
  Active involvement in recovery care services, including but not limited to Alcoholics Anonymous Narcotics Anonymous, individual counseling, methadone/suboxone program, etc. This information is obtained from self-report surveys administered by medical students in both conditions at both baseline and each follow-up.
Change in Substance Use Frequency | intervals of 1, 2, 3, and 6 months post-baseline assessment
  Frequency of substance use assessed using the 13-item Addiction Severity Index (ASI-Lite). The scale asks how many days in the last 30 days participants used each of several substances. The range of responses is 0 - 30 with higher scores indicating higher/greater severity of substance use.

SECONDARY OUTCOMES:
Change in Self-Reported Quality of Life Assessment | intervals of 1, 2, 3, and 6 months post-baseline assessment
  The 12-item Health-Related Quality of Life Short Form (SF-12) is used to obtain self-report information on participants' satisfaction with physical, psychological, social, and environmental aspects of their lives.Physical and Mental Health Composite Scores on the SF-12 are calculated using the score of all questions and range from 0 - 100. A zero score indicates the poor health and 100 indicates the highest level of health.

CONTACTS AND LOCATIONS:
Locations (1):
- Greenville Memorial Hospital, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cupp JA, Byrne KA, Herbert K, Roth PJ. Acute Care Utilization After Recovery Coaching Linkage During Substance-Related Inpatient Admission: Results of Two Randomized Controlled Trials. J Gen Intern Med. 2022 Aug;37(11):2768-2776. doi: 10.1007/s11606-021-07360-w. Epub 2022 Mar 16. PMID 35296984